CLINICAL TRIAL: NCT01696812
Title: Web-based International Multi-Center Clinical Study for Parkinson's Disease; the Evaluation of Clinical Outcome Based on the Electrode Position Estimated From the Fused Images of Preoperative MRI and Postoperative CT After Bilateral STN DBS
Brief Title: Web-based International Multi-Center Clinical Study for Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DELAS-201209; DELAS (Other Grant/Funding Number: H-1201-074-395)
Record Dates: First submitted 2012-09-18; First posted 2012-10-01 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2014-11

CONDITIONS: Parkinson Disease
Keywords: electrodeposition; Subthalamic Nucleus; Deep Brain Stimulation; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- electrode position, STN DBS, Parkinson' disease (Experimental): To determine the electrode positions with the relationship of the STN from the fused images of the preoperative MRI and the postoperative CT via web-site.
  Interventions: Procedure: electrode position

INTERVENTIONS:
Procedure: electrode position

SUMMARY:
The objectives of this study are (1) to compare the clinical outcome in correlation with the electrode positions estimated by web-based image fusion of the preoperative MRI and the postoperative brain CT taken at a stable period after surgery using mutual information technique in the patients with advanced Parkinson's disease (PD) after bilateral STN DBS and (2) to examine whether the documentation of the electrode position by using mutual information technique at a stable period after unilateral or bilateral STN stimulation provides useful information for the postoperative programming.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Parkinson Disease patients

Exclusion Criteria:

* The patients who have experienced any perioperative or postoperative complications
* The patients with severe cognitive impairment, ongoing psychiatric problems, an unsatisfactory general condition for evaluation, or an inability

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
To determine the electrode positions with the relationship of the STN from the fused images of the preoperative MRI and the postoperative CT | at 1 month after surgery

SECONDARY OUTCOMES:
UPDRS, H&Y, ADL scores, LEDD | at 6 and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sun Ha Paek, M.D., Ph.D., Principal Investigator — Department of Neurosurgery, Seoul National University Hospital
Locations (1):
- Department of Neurosurgery, Seoul National University Hospital, Seoul, Seoul, South Korea